CLINICAL TRIAL: NCT00315315
Title: A Prospective Study of Surgical Procedures for the Treatment of Persistent Nasolacrimal Duct Obstruction in Children Less Than Four Years Old
Brief Title: Study of Surgical Procedures for Treatment of Persistent Nasolacrimal Duct Obstruction in Children < 4 Years Old
Acronym: NLD2
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ray Kraker, Director, PEDIG Coordinating Center, Jaeb Center for Health Research
Other Study IDs: NEI-117; 2U10EY011751 (NIH); 5U10EY011751 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Nasolacrimal Duct Obstruction
Keywords: Nasolacrimal duct obstruction; Balloon catheter nasolacrimal duct dilation; Nasolacrimal intubation; Simple Nasolacrimal duct probing
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Nasolacrimal balloon catheter dilation — Balloon catheter nasolacrimal duct dilation consists of punctal dilation of at least one punctum and the passage into the nose of a semi-flexible wire probe with an inflatable balloon on the tip.
Procedure: Nasolacrimal intubation — Nasolacrimal duct intubation consists of punctal dilation of at least one punctum with the passage of a flexible lacrimal probe into the nose and the placement of a temporary stent in the nasolacrimal duct.
Procedure: Nasolacrimal duct probing — Simple nasolacrimal duct probing consists of punctal dilation of at least one punctum and the passage of a probe into the nose.

SUMMARY:
The purpose of this study is:

* To report the success proportions for the treatment of persistent nasolacrimal duct obstruction for three surgical procedures: balloon catheter dilation, nasolacrimal intubation, and simple probing.
* To obtain descriptive data regarding symptoms and quality of life in patients receiving each type of surgical procedure, and to compare success proportions between patients undergoing balloon catheter dilation and those undergoing nasolacrimal intubation.

DETAILED DESCRIPTION:
Nasolacrimal duct obstruction (NLDO) is a common ocular condition in the first year of life. As many as 95% of cases resolve spontaneously by one year of age. For those children in whom the condition does not resolve spontaneously, the initial surgical management is a probing of the nasolacrimal duct. Such a procedure is often successful, with cure rates up to 95%, especially in the first year of life. However, there are some patients in whom the initial procedure is not successful and repeat surgery is needed. Failure of an initial probing is thought to be associated with abnormal nasolacrimal anatomy, closure by healing of the surgical opening in the nasolacrimal duct, continued occlusion by the inferior turbinate, creation of a false passage, or faulty technique.

Several case series of repeat surgery for nasolacrimal obstruction have been reported. These studies have generally been retrospective, uncontrolled, unmasked, and conducted in single centers. These studies have also used differing definitions of treatment success, making it difficult to compare outcomes between the techniques. There is currently no accepted clinical practice for the management of these children. Clinicians choose among repeat probing, repeat probing with inferior turbinate infracture, multipass probing, balloon catheter dilation, and nasolacrimal duct intubation.

Repeat probing was for many years the only method available for persistent obstruction. However, because the repeat probing procedure was associated with failures, surgeons began to probe the nasolacrimal duct and to place a temporary stent in the nasolacrimal duct. Nasolacrimal duct intubation has been an alternative to probing for relief of NLDO for more than thirty years. Most often, silicone tubes are left in the drainage system for 1 to 3 months to allow time for complete healing around the tubes resulting in canalization. The stent is removed with topical anesthesia. Conscious sedation or general anesthesia may be utilized at investigator discretion. The reported success proportions for nasolacrimal intubation following failed probing vary from 69% to 100% in published reports.

More recently, the nasolacrimal probe has been combined with a balloon designed to forcibly expand the nasolacrimal duct, a strategy taken from angioplasty. The balloon catheter dilation has been available for the past 10 years. This procedure involves probing the nasolacrimal duct with a semi-flexible wire probe with an inflatable balloon on the tip. This technique has been used as a primary treatment of NLDO as well as a treatment for previous surgical failures. Balloon dilation has been promoted as a less complex procedure when compared to intubation, because it does not require retrieval of the probe from the nose. An additional advantage is that a stent is not left in the nasolacrimal system once the procedure is completed, eliminating the post-operative issues regarding removal of the tubes. The reported success proportions for balloon catheter dilation vary between 50% to 94% in published reports.

The public health importance of this study is the potential to reduce the total number of procedures necessary for NLDO after a failed probing as well as to reduce the need for dacryocystorhinostomy (DCR) surgery in children. Reductions in the number of these procedures will reduce health care expenditures and would be expected to be associated with a better quality of life for the patients.

The study has been designed as an observational study that largely approximates standard clinical practice. All procedures are consistent with standard care with the exception of a questionnaire which the patient's parent will complete at each study visit on NLDO symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - < 48 months
* Parent/guardian has the ability to complete a written questionnaire
* Onset of NLDO symptoms and/or signs prior to 6 months chronological age
* Presence of epiphora, increased tear film, and/or mucopurulent discharge in the absence of an upper respiratory infection or an ocular surface irritation
* Previous single failed simple probing procedure for nasolacrimal duct obstruction
* Investigator has determined the patient requires a second procedure for opening of the nasolacrimal duct

Exclusion Criteria:

* History of nasolacrimal intubation, balloon catheter dilation, more than one simple probing, or dacryocystorhinostomy
* Glaucoma present
* Corneal surface disease

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2005-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael X. Repka, M.D., Study Chair — Wilmer Eye Institute; David I. Silbert, M.D., Study Chair — Family Eye Group
Locations (2):
- United States (2):
  - Wilmer Eye Institute, Baltimore, Maryland
  - Family Eye Clinic, Lancaster, Pennsylvania

REFERENCES:
- [Result] Repka MX, Chandler DL, Holmes JM, Hoover DL, Morse CL, Schloff S, Silbert DI, Tien DR; Pediatric Eye Disease Investigator Group. Balloon catheter dilation and nasolacrimal duct intubation for treatment of nasolacrimal duct obstruction after failed probing. Arch Ophthalmol. 2009 May;127(5):633-9. doi: 10.1001/archophthalmol.2009.66. PMID 19433712